CLINICAL TRIAL: NCT01575366
Title: Movement Velocity Effect on Cortical Reorganization and Finger Function in Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0912M74993
Record Dates: First submitted 2012-03-19; First posted 2012-04-11 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow tracking training (Experimental)
  Interventions: Behavioral: Tracking training
- Fast tracking training (Experimental)
  Interventions: Behavioral: Tracking training

INTERVENTIONS:
Behavioral: Tracking training — The paretic finger movement training at different velocities included two 5-week periods of five days per week, 2-hours per day phases. The frequency for the higher-velocity training is 0.8 Hz, whereas the lower frequency training is 4 times slower, at 0.2 Hz. The two periods are each followed by a 3-week baseline period. The subject is seated in front of a laptop computer with the paretic forearm resting on the arm of the chair in a quiet room at home. The position of the forearm is pronated. An electrogoniometer, composed of a potentiometer attached to a custom hand splint, is placed on the paretic index finger with the potentiometer centered at the metacarpophalangeal joint. To keep the training session time equal between the two training phases, the duration of each slow training trial is 5 sec, compared to 20 sec for each fast training trial. Ultimately, the total number of required finger extension/flexion training movements is equal between the two phases.

SUMMARY:
Aim 1. Determine whether higher-velocity finger tracking training improves hand function more than slower velocity training. Working hypotheses: The higher-velocity training will have significantly greater functional improvement compared to the lower-velocity training, as measured by standardized upper extremity functional tests (Jebsen Taylor test, Box & Block Test, and Finger extension force test)

Aim 2. Ascertain whether higher-velocity finger tracking training differentially induces cortical reorganization as compared to lower-velocity finger tracking training.

Working hypotheses: The higher-velocity training will have significantly greater cortical reorganization compared to the lower-velocity training, as measured by:

1. TMS - increased amplitude of motor evoked potentials (MEP) from paretic extensor digitorum muscle in response to paired-pulse TMS to ipsilesional primary motor area (M1).
2. fMRI - increased volume of activation, signal intensity, and laterality of ipsilesional M1.

Aim 3. Explore whether the functional improvements correlate with the cortical reorganization. Working hypotheses: The functional improvements will correlate with the cortical reorganization.

ELIGIBILITY:
Inclusion criteria include:

* Ischemic stroke - due to higher risk of seizures in hemorrhagic stroke
* Subcortical location of stroke
* Stroke after 6 months - lower limit of 6 months to avoid confounding from spontaneous recovery (Jorgensen, Nakayama et al. 1995) and no upper limit to maximize pool of candidate subjects while still showing training effect (Carey, Kimberley et al. 2002)
* At least 18 years of age - to maximize pool of candidate subjects
* Mini-Mental State Examination score >24 - to ensure satisfactory cognition to perform tasks
* Satisfactory corrected vision - to see computer screen during training and testing
* Active range of MP joint at paretic index finger of at least 10 degrees - based on minimal movement required to perform training task successfully, and that larger amplitudes would reduce the pool of subjects available for participating in the study.
* Ability to pronate the forearm so that index finger extension movement during training is vertically upward and relaxation results in the finger falling back to the flexed starting position
* not currently receiving any other therapy - to avoid confounding treatment effects
* Approval for participation by a neurologist - to ensure subject is reasonably safe to receive TMS testing. Subjects with proprioceptive loss or expressive aphasia will be included, providing they can carryout the training task.

Exclusion criteria include:

* Inability to follow 3-step commands
* A visual field cut that causes subjects not to see all indicators on a computer screen positioned centrally in from of them
* History of seizures
* Family member with history of seizures
* Presence of any other neuromuscular disorders
* Pregnancy
* Claustrophobia
* Indwelling metal or medical devices/implants incompatible with functional fMRI testing
* History of exposure to finger tracking training.
* Informed consent will be obtained and TMS/fMRI safety screenings will be conducted prior to testing procedures.
* Subjects will be recruited as volunteers from letters sent to previous research subjects inviting their participation, through visits to local stroke support groups meetings, newspaper advertisements and referrals from neurologists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Hand function improvement | taken at weekly intervals for the whole study length, 20 weeks.
  Jebsen Taylor test, Box & Block Test, and Finger extension force test

SECONDARY OUTCOMES:
corticospinal excitability | taken at weekly intervals for the whole study length, 20 weeks.
  TMS
cognitive function | at the beginning and at the end of the study, which are 1st and 20th week.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiong Deng, MD, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States